CLINICAL TRIAL: NCT04970316
Title: Organ Specific Late Adverse Effects, in Colorectal Cancer Patients Following Surgery With Either HIPEC or Pelvic Exenteration
Brief Title: Late Organ Specific Adverse Effects hiPec or pElvic eXenteration
Acronym: LOSAPEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Karolinska University Hospital (Other); Skane University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LOSAPEX
Record Dates: First submitted 2021-06-28; First posted 2021-07-21 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer
Keywords: cytoreductive surgery; hyperthermic intraperitoneal chemotherapy; pelvic exenteration; adverse effects; bowel dysfunction; urinary dysfunction; sexual dysfunction; pain; lymphedema
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Diseases; Sexual Dysfunction, Physiological; Pain; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIPEC cohort: Patients undergoing cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) for colorectal cancer with peritoneal metastases
- PE cohort: Patients undergoing pelvic exenteration (PE) for colorectal cancer with involvement of the urinary bladder

SUMMARY:
The purpose of this study is to describe type and extent of organ specific late adverse effects in patients undergoing surgery for colorectal cancer with peritoneal metastases and after surgery for colorectal cancer with involvement of the urinary bladder.

DETAILED DESCRIPTION:
After being informed about the study all patients giving written informed consent will be distributed a questionnaire asking questions on bowel function, urinary function, pain, sexual function and lymphedema. All these aspects will be investigated using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone intended curative CRS+HIPEC for peritoneal metastases originated from colorectal cancer (HIPEC cohort) according to national Danish guidelines
* Patients who have undergone intended curative total or anterior pelvic exenteration (PE cohort) for advanced or recurrent colorectal cancer according to national Danish guidelines

Exclusion Criteria:

* Patients under 18 years
* Patients not speaking Danish or Swedish, respectively, in Denmark and Sweden
* Patients unable to give informed consent
* Patients undergoing CRS+HIPEC or PE for cancers others than CRC
* Terminally ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will prospectively include patients who have undergone surgery at Aarhus University Hospital, Karolinska University Hospital, Stockholm, and Skåne University Hospital, Malmö. Inclusion in Denmark will start February 2021 and in Sweden Summer 2021. Inclusion period is 15 months.
  The HIPEC cohort will be established as a cross-sectional study. For newly operated patients, inclusion will happen shortly after surgery with prospective questionnaire follow-ups at 3, 6 and 12 months after inclusion. For patients who have undergone CRS+HIPEC more than 3 months ago, initial inclusion can take place at 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Patients in the PE cohort will be included shortly after surgery with follow-up at 3 months, 6 months and 12 months after surgery.
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Development of bowel related adverse effects after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionnaires: Skt. Marks incontinence score
Development of bowel related adverse effects after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionnaires: Wexner incontinence score
Development of bowel related adverse effects after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionnaires: LARS score (low anterior resection syndrome)
Development of male urological dysfunction after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionaires: ICIQ-MLUTS (ICIQ male lower urinary tract symptoms)
Development of female urological dysfunction after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionaires: ICIQ-FLUTS (ICIQ female lower urinary tract symptoms)
Development of male sexual dysfunction after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionaires: IIEF-5 (international index of erectile dysfunction)
Development of female sexual dysfunction after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionaires: Rectal cancer female sexuality score
Development of pain after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionaire: rectal cancer pain score
Development of lymphedema after PE for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery
  Descriptive analysis will be done using following questionaire: Questions regarding lymphedema from EORTC vulva cancer questionnaire
Development of stoma-related issues after PE or CRS+HIPEC for colorectal cancer | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects 3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Descriptive analysis will be done using following questionaire: Colostomy impact score

SECONDARY OUTCOMES:
Risk factors associated with developing organ specific late adverse effects | PE cohort: Development and change in adverse effects 3, 6 and 12 months after surgery. HIPEC cohort: Development and change in adverse effects3, 6, 12, 18, 24, 36, 48 and 60 months after surgery.
  Univariate and multivariate regression analysis will be performed to identify potential risk factors for developing these adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Rogini Balachandran, MD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Department of Surgery, Aarhus University Hospital, Aarhus, Denmark
- Sweden (2):
  - Department of Surgery, Karolinska University Hospital, Solna, Stockholm County
  - Department of Surgery, Skånes University Hospital, Malmö, Malmo

IPD SHARING:
Plan to Share IPD: No